CLINICAL TRIAL: NCT02748421
Title: Evaluation Use Optical Coherence Tomography - Rescan During Dissection of Macular Membranes : Pre and Post Operative Aspects
Brief Title: Optical Coherence Tomography - Rescan During Dissection of Macular Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Instituto Paulista de Estudos e Pesquisa em Oftalmologia (Other)
Responsible Party: Principal Investigator, Michel Eid Farah, Michel Eid Farah, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 50991615.6.0000.5505
Record Dates: First submitted 2016-04-06; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Macular Hole; Epiretinal Membrane; Traction Syndrome Vitreomacular; Proliferative Vitreoretinopathy
Keywords: retina surgery; image guided surgery; optical coherence tomography assisted
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane; Vitreoretinopathy, Proliferative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumera Microscope with OCT RESCAN (Other): in the group microscope coupled to OCT, patients will undergo retinal surgery using the Lumera microscope with Rescan OCT Zeiss
  Interventions: Procedure: Lumera Microscope with OCT RESCAN
- Conventional Microscope (Other): control group without OCT RESCAN
  Interventions: Procedure: Conventional Microscope

INTERVENTIONS:
Procedure: Lumera Microscope with OCT RESCAN — macular membrane dissection with OCT RESCAN
  Arms: Lumera Microscope with OCT RESCAN
Procedure: Conventional Microscope — macular membrane dissection without OCT RESCAN
  Arms: Conventional Microscope

SUMMARY:
In our study , the investigators will use the microscope with OCT ( Lumera with RESCAN OCT ) coupled to assess the extent , depth and change of retinal architecture in the perioperative period . Thus , they will evaluate what the optimal maneuvers of dissection of macular membranes to obtain a more satisfactory result of the rearrangement in the retinal layers . Furthermore , the use of OCT perioperative may dispense with the use of dyes , decreasing the concentration used or reduce the exposure time. Thus, they can get the potential decrease in retinal toxicity may be generated by them.

DETAILED DESCRIPTION:
The investigators will use the microscope with OCT (Lumera with RESCAN OCT) coupled to assess the extent, depth and change of retinal architecture in the perioperative period. Thus, they will evaluate what the optimal maneuvers of dissection of macular membranes to obtain a more satisfactory result of the rearrangement in the retinal layers. Furthermore, the use of OCT perioperative may dispense with the use of dyes, decreasing the concentration used or reduce the exposure time.

Materials and methods The investigators will evaluate 30 patients with changes in macular membranes with surgical removal of indication from the Retina and Vitreous outpatient sector of Unifesp - Paulista School of Medicine. The patients will be classified according to the diseases in the following groups: Macular Hole, Epiretinal Membrane, Traction Syndrome vitreomacular, and proliferative vitreoretinopathy of Retinal Detachment. Everyone will be informed about the risks and benefits of the study and sign an informed consent form. In the preoperative evaluation a complete ophthalmologic examination with complementary tests such as angiography and optical coherence tomography will be done.

Patients will undergo retinal surgery using the Lumera Microscope WITH RESCAN OCT - ZEISS. The team of surgeons will answer the questionnaire on the surgical difficulty regarding the identification and removal of macular membranes.

All patients will be assessed at 1, 7, 15, 30, 60 and 90 and 180 days after surgery, including the following tests:

* Measurement of visual acuity with best correction
* Previous Biomicroscopy
* Indirect Funduscopy
* tonometry
* Optical coherence tomography (OCT)
* Retinography Surgeries and procedures of the study groups will be conducted by the same team of surgeons and all surgeries and procedures will be carried out in IPEPO - Paulista Institute of Studies and Research in Ophthalmology / Vision Institute.

For each type of retinal disease, there will be a control group and a group OCT as detailed below: 1 - GROUP CONTROL The control group will undergo retinal surgery with conventional microscope without coupled OCT. This group will have its filmed and documented surgery. The team of surgeons will answer the questionnaire on the surgical difficulty regarding the identification and removal of macular membranes.

2 -GROUP OCT / RESCAN In the group microscope coupled to OCT, patients will undergo retinal surgery using the Lumera Microscope WITH RESCAN OCT - ZEISS and have their filmed and documented surgery. The team of surgeons will answer the questionnaire on the surgical difficulty regarding the identification and removal of macular membranes.

Statistical methodology All information will be presented by mean and standard deviation for the quantitative variables and absolute frequency (n) and relative (%) for qualitative variables.

ELIGIBILITY:
Inclusion criteria:

* Visual acuity less than 20/60 in the affected eye
* 18 years of both sexes
* 1 diagnostics of the diseases Macular Hole,Epiretinal membrane,Traction Syndrome vitreomacular, vitreoretinopathy Proliferative Retina Detachment.
* Indication of vitreoretinal surgery

Exclusion criteria:

* Any previous eye surgery in the study eye
* Better visual acuity than or equal to 20/60.
* Any previous infection affecting any eye structure. transport costs and feeding of patients will be the responsibility of the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Assess optimal maneuvers in macular membrane dissection | Day 0 (surgical day)
  by a questionnaire responded by surgeons (no difficulty, some difficulty, very difficulty)

SECONDARY OUTCOMES:
Compare the time of surgery between groups | Day 0 (surgical day)
  by a questionnaire responded by surgeons (until 1 hour, between 1-2 hours, more than 2 hours
describe the surgical difficulty for macular membrane dissection | Day 0
  by a questionnaire responded by surgeons (no difficulty, some difficulty, very difficulty)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Farah, MD, PhD, Principal Investigator — Federal University of São Paulo UNIFESP

IPD SHARING:
Plan to Share IPD: Yes
scientific publication